CLINICAL TRIAL: NCT06330064
Title: A Phase 1B/2 Pan-Tumor, Open-Label Study To Evaluate The Efficacy And Safety Of Ifinatamab Deruxtecan (I-DXd) In Subjects With Recurrent Or Metastatic Solid Tumors (IDeate-PanTumor02)
Brief Title: A Study To Evaluate The Efficacy And Safety Of Ifinatamab Deruxtecan (I-DXd) In Subjects With Recurrent Or Metastatic Solid Tumors (IDeate-PanTumor02)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DS7300-203; 2023-509632-26-00 (Other: EU CTR); JRCT2031240016 (Other: JRCT)
Record Dates: First submitted 2024-03-19; First posted 2024-03-26 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Recurrent or Metastatic Solid Tumors
Keywords: Recurrent or metastatic solid tumors; Endometrial cancer; Head and neck squamous cell carcinoma; Colorectal cancer; Hepatocellular carcinoma; Adenocarcinoma of esophagus, gastroesophageal junction, and stomach; Urothelial carcinoma; Ovarian cancer; Cervical cancer; Biliary tract cancer; Human epidermal growth factor 2 (HER2)-low breast cancer; HER2 immunohistochemistry 0 breast cancer; Cutaneous melanoma; Pancreatic ductal adenocarcinoma; Ifinatamab deruxtecan (I-DXD); DS7300a
MeSH Terms: conditions — Recurrence; Endometrial Neoplasms; Squamous Cell Carcinoma of Head and Neck; Colorectal Neoplasms; Carcinoma, Hepatocellular; Adenocarcinoma Of Esophagus; Carcinoma, Transitional Cell; Ovarian Neoplasms; Uterine Cervical Neoplasms; Biliary Tract Neoplasms; Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (13):
- Cohort 1: Endometrial Cancer (Experimental): Participants with recurrent or metastatic endometrial cancer who were previously treated with 1 or more systemic therapy who received an intravenous infusion of I-DXd 12 mg/kg.
  Interventions: Drug: Ifinatamab deruxtecan
- Cohort 2: Head and Neck Squamous Cell Carcinoma (Experimental): Participants with recurrent or metastatic head and neck squamous carcinoma who were previously treated with 1 or more systemic therapy who received an intravenous infusion of I-DXd 12 mg/kg.
  Interventions: Drug: Ifinatamab deruxtecan
- Cohort 3: Pancreatic Ductal Adenocarcinoma (Experimental): Participants with recurrent or metastatic pancreatic ductal adenocarcinoma who were previously treated with 1 or more systemic therapy who received an intravenous infusion of I-DXd 12 mg/kg.
  Interventions: Drug: Ifinatamab deruxtecan
- Cohort 4: Colorectal Cancer (Experimental): Participants with recurrent or metastatic colorectal cancer who were previously treated with 1 or more systemic therapy who received an intravenous infusion of I-DXd 12 mg/kg.
  Interventions: Drug: Ifinatamab deruxtecan
- Cohort 5: Hepatocellular Carcinoma (Experimental): Participants with recurrent or metastatic hepatocellular carcinoma who were previously treated with 1 or more systemic therapy who received an intravenous infusion of I-DXd at the determined dose.
  Interventions: Drug: Ifinatamab deruxtecan
- Cohort 6: Adenocarcinoma of esophagus, gastroesophageal junction, and stomach (Experimental): Participants with recurrent or metastatic adenocarcinoma of esophagus, gastroesophageal junction, and stomach who were previously treated with 1 or more systemic therapy who received an intravenous infusion of I-DXd 12 mg/kg.
  Interventions: Drug: Ifinatamab deruxtecan
- Cohort 7: Urothelial carcinoma (Experimental): Participants with recurrent or metastatic urothelial carcinoma who were previously treated with 1 or more systemic therapy who received an intravenous infusion of I-DXd 12 mg/kg.
  Interventions: Drug: Ifinatamab deruxtecan
- Cohort 8: Ovarian cancer (Experimental): Participants with recurrent or metastatic non-squamous ovarian cancer who were previously treated with 1 or more systemic therapy who received an intravenous infusion of I-DXd 12 mg/kg.
  Interventions: Drug: Ifinatamab deruxtecan
- Cohort 9: Cervical cancer (Experimental): Participants with recurrent or metastatic cervical cancer who were previously treated with 1 or more systemic therapy who received an intravenous infusion of I-DXd 12 mg/kg.
  Interventions: Drug: Ifinatamab deruxtecan
- Cohort 10: Biliary tract cancer (Experimental): Participants with recurrent or metastatic biliary tract cancer who were previously treated with 1 or more systemic therapy who received an intravenous infusion of I-DXd 12 mg/kg.
  Interventions: Drug: Ifinatamab deruxtecan
- Cohort 11: Human epidermal growth factor 2 (HER2)-low breast cancer (Experimental): Participants with recurrent or metastatic human epidermal growth factor 2 (HER2)-low breast cancer who were previously treated with 1 or more systemic therapy who received an intravenous infusion of I-DXd 12 mg/kg.
  Interventions: Drug: Ifinatamab deruxtecan
- Cohort 12: HER2 immunohistochemistry (IHC) 0 breast cancer (Experimental): Participants with recurrent or metastatic HER2 immunohistochemistry (IHC) 0 breast cancer who were previously treated with 1 or more systemic therapy who received an intravenous infusion of I-DXd 12 mg/kg.
  Interventions: Drug: Ifinatamab deruxtecan
- Cohort 13: Cutaneous melanoma (Experimental): Participants with recurrent or metastatic cutaneous melanoma who were previously treated with 1 or more systemic therapy who received an intravenous infusion of I-DXd 12 mg/kg.
  Interventions: Drug: Ifinatamab deruxtecan

INTERVENTIONS:
Drug: Ifinatamab deruxtecan — Intravenous administration
  Other Names: I-DXd

SUMMARY:
This study is designed to assess the efficacy and safety of ifinatamab deruxtecan (I-DXD) in the following tumor types: endometrial cancer (EC); head and neck squamous cell carcinoma (HNSCC); pancreatic ductal adenocarcinoma (PDAC); colorectal cancer (CRC); hepatocellular carcinoma (HCC); adenocarcinoma of esophagus, gastroesophageal junction, and stomach (Ad-Eso/GEJ/gastric); urothelial carcinoma (UC); ovarian cancer (OVC); cervical cancer (CC); biliary tract cancer (BTC); human epidermal growth factor 2 (HER2)-low breast cancer (BC); HER2 immunohistochemistry (IHC) 0 BC; and cutaneous melanoma.

DETAILED DESCRIPTION:
This study will evaluate the efficacy and safety of I-DXd in participants with recurrent or metastatic solid tumors previously treated with 1 or more systemic therapies for the selected tumor indication. The study will be divided into 2 parts: Stage 1 and Stage 2. Each cohort starts with Stage 1 and may continue to Stage 2 if sufficient safety and efficacy data are observed.

The HCC Safety Run-In (Phase 1) will assess the safety and tolerability of I-DXd in participants with HCC.

ELIGIBILITY:
Participants must meet all of the following criteria to be included in the study:

Common Inclusion Criteria for All Participants

1. Participant must have at least 1 lesion, not previously irradiated, amenable to core biopsy and must consent to provide a pretreatment biopsy tissue sample. An archival tumor tissue sample obtained within 6 months of consent and after progression during/after treatment with the participant's most recent cancer therapy regimen is also acceptable.
2. Participants ages ≥18 years (follow local regulatory requirements if the legal age of consent for study participation is >18 years).
3. At least 1 measurable lesion on computed tomography (CT) or magnetic resonance imaging (MRI) according to Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1), as assessed by the investigator.
4. Documentation of radiological disease progression on or after the previous standard-of-care regimen in the advanced/metastatic setting.
5. Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.

Additional Inclusion Criteria for EC Participants

1. Pathologically or cytologically documented EC of any histological carcinoma subtype or endometrial carcinosarcoma, irrespective of microsatellite instability or mismatch repair status.
2. Relapse or progression after a platinum-containing systemic treatment and an immune checkpoint inhibitor (ICI)-containing regimen (combined or sequential). Subjects with actionable target tumor mutation should have been previously treated with targeted therapy, with a maximum of 3 prior lines of therapy for endometrial carcinoma or carcinosarcoma. Neoadjuvant/adjuvant therapy may count as 1 line of therapy if the subject progressed within 6 months after completion of therapy.

Additional Inclusion Criteria for HNSCC Participants

1. Pathologically or cytologically documented unresectable or metastatic squamous cell carcinoma of the oral cavity, oropharynx, hypopharynx, or larynx, excluding nasopharynx, nasal cavity and paranasal sinuses, and unknown primary.
2. Has disease progression after platinum-based and ICI treatment, whether administered in combination or separately. Subjects with actionable target tumor mutation should have been previously treated with targeted therapy, with a maximum of 2 prior therapy lines for unresectable or metastatic HNSCC.
3. Participants without radiographic evidence of major blood vessel invasion/infiltration or tumor demonstrating a >90-degree abutment or encasement of a major blood vessel.
4. Participants with no prior history of Grade ≥3 bleeding as per the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) v5.0 within 28 days prior to the start of study drug related to the current head and neck cancer may be included in the study.
5. Documented p16 status for oropharyngeal cancer (historical results are acceptable if available).

Additional Inclusion Criterion for PDAC Participants

1. Pathologically or cytologically documented unresectable or metastatic pancreatic adenocarcinoma that has relapsed or progressed after 1 prior line of gemcitabine-based systemic therapy in the locally advanced/metastatic setting or after 2 lines of therapy if the subject has actionable target tumor mutation and has been previously treated with targeted therapy. No prior treatment with topoisomerase I inhibitors, such as irinotecan or topotecan.

Additional Inclusion Criteria for CRC Participants

1. Pathologically or cytologically documented unresectable or metastatic CRC with microsatellite stable status.
2. Relapse or progression after 1 prior line of systemic therapy including a fluoropyrimidine plus oxaliplatin with or without anti-vascular endothelial growth factor (VEGF) monoclonal antibody (mAb) or anti-epidermal growth factor receptor mAb therapy, as clinically indicated, or relapse or progression after 2 lines of therapy if the subject has received targeted therapy.

   Note: Prior adjuvant/neoadjuvant systemic cytotoxic chemotherapy will count as 1 line of prior systemic therapy if there is documented disease progression during therapy or within 6 months of chemotherapy completion.
3. No prior treatment with topoisomerase I inhibitors, such as irinotecan or topotecan.

Additional Inclusion Criteria for HCC Participants

1. Pathologically or cytologically documented unresectable or metastatic HCC (fibrolamellar and mixed hepatocellular/cholangiocarcinoma subtypes are not eligible) or noninvasive diagnosis of HCC as per the American Association for the Study of Liver Diseases (AASLD) criteria in subjects with a confirmed diagnosis of cirrhosis.
2. Relapse or progression after 1 prior line of an ICI-containing regimen (combination or monotherapy) in the locally advanced/metastatic setting, with a maximum of 2 prior lines. Subjects with actionable target tumor mutation should have been previously treated with targeted therapy.
3. Barcelona Clinic Liver Cancer (BCLC) Stage B or C.
4. Liver function status should be Child-Pugh (CP) Class A.
5. Albumin-Bilirubin (ALBI) Grade 1 within 7 days prior to the first dose of study drug.
6. Participants with large esophageal varices at risk of bleeding must be treated with conventional medical intervention: beta blockers or endoscopic treatment.

Additional Inclusion Criteria for Ad-eso/GEJ/Gastric Participants

1. Pathologically or cytologically documented unresectable or metastatic Ad-eso/GEJ/Gastric that has relapsed or progressed after 1 prior line of systemic therapy in the locally advanced/metastatic setting. Subjects with PD-(L)1+ or MSI-H/dMMR should receive ICI treatment if ICIs are standard of care in the country, unless the subject is ineligible for ICI treatment.
2. If the participant has known history of HER2 positivity (defined by IHC 3+ or IHC 2+ and in situ hybridization [ISH] positive, as classified by American Society of Clinical Oncology - College of American Pathologists [ASCO CAP]) or actionable target, the subject must have been previously treated with a targeted therapy.

Additional Inclusion Criteria for UC Participants

1. Pathologically or cytologically documented unresectable or metastatic UC of the bladder, renal pelvis, ureter, or urethra. Participants with histological variants are allowed if urothelial histology is predominant. Small cell/neuroendocrine tumors are not allowed even if mixed histology.
2. Relapse or progression after at least 1 prior line of ICI-containing systemic therapy, and 1 prior line of systemic chemotherapy, given in combination with other anticancer therapy or separately, with a maximum of 3 prior therapy lines.

   1. At least 1 line of therapy should include enfortumab vedotin in countries where enfortumab vedotin is approved and available.
   2. Perioperative systemic therapies will be counted as 1 line of therapy.
   3. To meet inclusion criteria requirement of prior ICI-containing therapy, use in the perioperative or metastatic setting will suffice.
   4. Subjects with actionable target tumor mutation should have been previously treated with targeted therapy.
   5. The same regimen administered twice in different disease settings will be counted as 1 line of prior therapy.

Additional Inclusion Criteria for CC Participants

1. Histologically confirmed unresectable or metastatic CC that was previously treated with ≥1 prior line of systemic therapy in the locally advanced or metastatic setting. Subjects with actionable target tumor mutation should have been previously treated with targeted therapy.
2. Participants should receive prior anti-programmed death 1/programmed death-ligand 1 treatment and/or tisotumab vedotin if those are standard of care in the country, unless the subject is ineligible for these treatments.

Additional Inclusion Criteria for OVC Participants

1. Histologically confirmed high-grade serous OVC, high-grade endometrioid OVC, primary peritoneal cancer, or fallopian tube cancer that was previously treated with at least 1 line of platinum-based therapy and bevacizumab unless the subject is ineligible for treatment with bevacizumab.
2. Participant is no longer considered eligible for platinum-based therapy per the investigator's opinion or has progressed less than 180 days after the last dose of platinum therapy.
3. Participant is not considered primary platinum refractory and has not progressed during platinum treatment or within 4 weeks after the completion of platinum treatment.
4. Subjects with actionable target tumor mutation should have been previously treated with targeted therapy.

Additional Inclusion Criteria for BTC Participants

1. Pathologically or cytologically documented unresectable or metastatic BTC (intra- or extrahepatic cholangiocarcinoma or gallbladder carcinoma).
2. Relapse or progression after at least 1 prior line of systemic therapy, or 2 prior lines of systemic therapy if the participant has an actionable target and has received targeted therapy.
3. Histological subtypes other than ampullary cancer, small cell cancer, lymphoma, sarcoma, neuroendocrine tumors, mixed tumor histology, and/or mucinous cystic neoplasms (Please note that the histological subtypes listed here are not allowed.)

Additional Inclusion Criteria for HER2-Low BC Participants

1. Pathologically or cytologically documented unresectable or metastatic BC.
2. Low HER2 expression, defined as IHC 2+/ISH- or IHC 1+ (ISH- or untested), according to ASCO-CAP 2018 HER2 testing guidelines, based on most recent testing, regardless of hormonal status.
3. Progression on or after treatment with trastuzumab deruxtecan (T-DXd).
4. Relapse or progression after at least 2 and a maximum of 3 prior lines of systemic therapy. Subjects with metastatic hormone receptor (HR)+ BC who have received endocrine-based therapy and have received at least 2 and a maximum of 3 prior lines of additional systemic therapy in the metastatic setting. Subjects with actionable target tumor mutation should have been previously treated with targeted therapy.

Additional Inclusion Criteria for HER2 IHC 0 BC Participants

1. Pathologically or cytologically documented unresectable or metastatic BC.
2. Negative for HER2 expression, defined as IHC 0 (ISH- or untested) according to ASCO-CAP 2018 HER2 testing guidelines, based on the most recent testing, regardless of hormonal status.
3. Relapse or progression after at least 2 and a maximum of 3 prior lines of systemic therapy. Participants with metastatic HR+ BC who have received endocrine-based therapy and have received at least 2 and a maximum of 3 prior lines of additional systemic therapy in the metastatic setting. Subjects with actionable target tumor mutation should have been previously treated with targeted therapy.

Additional Inclusion Criteria for Cutaneous (Acral and Non-acral) Melanoma Subjects

1. Histologically or cytologically confirmed cutaneous (acral and non-acral) melanoma.
2. Disease progression while on or after having received treatment with ≥1 prior line of ICI based therapy. Prior anti-PD-(L)1 therapy in the adjuvant setting may be counted as 1 line if there is recurrence within 12 weeks of the last dose. If the subject had BRAF mutated melanoma or other actionable target tumor mutation, they must have had disease progression on targeted therapy as well.

Participants who meet any of the following criteria will be disqualified from entering the study:

1. Prior treatment with orlotamab, enoblituzumab, or other B7-homologue 3 (B7-H3)-targeted agents, including I-DXd.
2. Prior discontinuation of an antibody drug conjugate (ADC) that consists of an exatecan derivative (eg, T-DXd) due to treatment-related toxicities.
3. Clinically active brain metastases, spinal cord compression, or leptomeningeal carcinomatosis, defined as untreated or symptomatic, or requiring therapy with steroids or anticonvulsants to control associated symptoms.
4. Inadequate treatment washout period before enrollment as specified in the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 520 (Estimated)
Dates: Start 2024-04-10 (Actual); Primary Completion 2028-07-25 (Estimated); Study Completion 2028-07-25 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) as Assessed by Investigator | From the time of the first dose of study drug until the date of documented disease progression, death, loss to follow-up, or withdrawal by the subject, whichever occurs first up to approximately 57 months
  ORR is defined as the proportion of participants with a best overall response (BOR) of confirmed complete response (CR) or confirmed partial response (PR) as assessed by Investigator per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.
Number of Participants Reporting Dose-limiting Toxicities in the HCC Cohort | Cycle 1 Day 1 to Cycle 1 Day 21
  A dose-limiting toxicity (DLT) is defined as any treatment-emergent adverse event (TEAE) not attributable to disease or disease-related processes that occurs during the DLT evaluation period (from C1D1 to the end of Cycle 1 in Safety Run-in) and is Grade 3 or above, according to NCI-CTCAE version 5.0, with the exceptions as noted in the protocol.
Number of Participants Reporting Treatment-emergent Adverse Events and Death in the HCC Cohort | From date of signing the informed consent form up to 47 days after the last dose of study drug , up to approximately 57 months
  A TEAE is defined as an adverse event (AE) with a start or worsening date during the on-treatment period. AEs will be coded using MedDRA and will be graded using NCI-CTCAE v5.0.

SECONDARY OUTCOMES:
Incidence of Treatment Emergent Adverse Events (TEAEs), Serious Adverse Events (SAEs), and Adverse Events of Special Interest (AESIs) | From date of signing the informed consent form up to 47 days after the last dose of study drug , up to approximately 57 months
  A TEAE is defined as an adverse event (AE) with a start or worsening date during the on-treatment period. A serious AE is defined as any untoward medical occurrence that at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, is an important medical event, or may jeopardize the participant or may require medical or surgical intervention to prevent one of the other outcomes noted. AESIs will also be assessed. AEs will be coded using MedDRA and will be graded using NCI-CTCAE v5.0.
Duration of Response (DoR) | From the time of the first dose of study drug until the date of documented disease progression (confirmed by investigator), death, loss to follow-up, or withdrawal by the subject, whichever occurs first, up to approximately 57 months
  DoR is defined as the time from the first documented confirmed response (CR or PR) to the date of progression or death due to any cause as assessed by Investigator per RECIST v1.1, respectively. CR was defined as a disappearance of all target and non-target lesions and PR was defined as at least a 30% decrease in the sum of diameters of target lesions.
Progression-free Survival (PFS) | From the time of the first dose of study drug until the date of documented disease progression, death, loss to follow-up, or withdrawal by the subject, whichever occurs first, up to approximately 57 months
  PFS is defined as the time from the start of study treatment to the earlier of the dates of the first documentation of objective progressive disease (PD) per RECIST v1.1 or death due to any cause. PFS will be determined by the Investigator.
Disease Control Rate (DCR) | From the time of the first dose of study drug until the date of documented disease progression (by investigator), death, loss to follow-up, or withdrawal by the subject, whichever occurs first, up to approximately 57 months
  DCR is defined as the proportion of participants who achieved a BOR of confirmed CR, confirmed PR, or stable disease (SD) as assessed by the Investigator per RECIST v1.1, respectively. CR was defined as a disappearance of all target and non-target lesions, PR was defined as at least a 30% decrease in the sum of diameters of target lesions, and stable disease (SD) was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD; at least a 20% increase in the sum of diameters of target lesions.
Overall Survival (OS) | From the date of the first dose of drug up to the date of death due to any cause, up to approximately 57 months
  OS is defined as the time interval from the date of the first dose of study drug to the date of death from any cause.
Pharmacokinetic Parameter Maximum Concentration (CMax) for I DXd, total anti-B7-H3 antibody, and DXd | Cycles 1 and 3 Day 1: predose, end of infusion, 3 hours (hr), 6 hr; 24 hr, 168 hr; 336 hr; 504 hr; Cycles 2, 4, and 5 Day 1: predose and end of infusion; Cycle 7 and every 2 cycles thereafter up to EOS (57 months) predose (every cycle is 21 days)
  Plasma pharmacokinetic parameters will be estimated using noncompartmental methods.
Pharmacokinetic Parameter Time to Reach Maximum Plasma Concentration (TMax) for I DXd, total anti-B7-H3 antibody, and DXd | Cycles 1 and 3 Day 1: predose, end of infusion, 3 hours (hr), 6 hr; 24 hr, 168 hr; 336 hr; 504 hr; Cycles 2, 4, and 5 Day 1: predose and end of infusion; Cycle 7 and every 2 cycles thereafter up to EOS (57 months) predose (every cycle is 21 days)
  Plasma pharmacokinetic parameters will be estimated using noncompartmental methods.
Pharmacokinetic Parameter Half-life (t1/2) for I DXd, total anti-B7-H3 antibody, and DXd | Cycles 1 and 3 Day 1: predose, end of infusion, 3 hours (hr), 6 hr; 24 hr, 168 hr; 336 hr; 504 hr; Cycles 2, 4, and 5 Day 1: predose and end of infusion; Cycle 7 and every 2 cycles thereafter up to EOS (57 months) predose (every cycle is 21 days)
  Plasma pharmacokinetic parameters will be estimated using noncompartmental methods.
Pharmacokinetic Parameter Minimum Concentration (Ctrough) for I DXd, total anti-B7-H3 antibody, and DXd | Cycles 1 and 3 Day 1: predose, end of infusion, 3 hours (hr), 6 hr; 24 hr, 168 hr; 336 hr; 504 hr; Cycles 2, 4, and 5 Day 1: predose and end of infusion; Cycle 7 and every 2 cycles thereafter up to EOS (57 months) predose (every cycle is 21 days)
  Plasma pharmacokinetic parameters will be estimated using noncompartmental methods.
Pharmacokinetic Parameter Area Under the Curve (AUC) for I DXd, total anti-B7-H3 antibody, and DXd | Cycles 1 and 3 Day 1: predose, end of infusion, 3 hours (hr), 6 hr; 24 hr, 168 hr; 336 hr; 504 hr; Cycles 2, 4, and 5 Day 1: predose and end of infusion; Cycle 7 and every 2 cycles thereafter up to EOS (57 months) predose (every cycle is 21 days)
  Plasma pharmacokinetic parameters will be estimated using noncompartmental methods.
Percentage of Participants Who Are Anti-Drug Antibody (ADA)-Positive (Baseline and Post-Baseline) | Baseline up to 57 months
  Anti-drug antibodies will be measured in the plasma using a validated assay.
Percentage of Participants Who Have Treatment-emergent ADA | Baseline up to 57 months
  Anti-drug antibodies will be measured in the plasma using a validated assay.

CONTACTS AND LOCATIONS:
Locations (118):
- United States (17):
  - Los Angeles Cancer Network, Los Angeles, California
  - Valkyrie Clinical Trials, Los Angeles, California
  - Pih Health Hematology Medical Oncology, Whittier, California
  - Orchard Healthcare Research Inc., Skokie, Illinois
  - M Health Fairview University of Minnesota Medical Center, Minneapolis, Minnesota
  - NYU Langone Health, New York, New York
  - Icahn School of Medicine At Mount Sinai Prime, New York, New York
  - Clinical Research Alliance, Westbury, New York
  - Tn Gynecologic Oncology Group, Llc, Chattanooga, Tennessee
  - The West Clinic, Germantown, Tennessee
  - SCRI Oncology Partners, Nashville, Tennessee
  - Texas Oncology - West Texas, Amarillo, Texas
  - Texas Oncology, P.A., Dallas, Texas
  - Texas Oncology Gulf Coast, Pearland, Texas
  - University of Utah Hospitals & Clinics, Salt Lake City, Utah
  - Virginia Cancer Specialists, Fairfax, Virginia
  - Wenatchee Hospitals and Clinics, Wenatchee, Washington
- Argentina (5):
  - DIABAID, Buenos Aires
  - Hospital Aleman, Buenos Aires
  - Hospital Sirio Libanes, Caba
  - Centro Médico Austral, Ciudad Autonoma Buenos Aires
  - Centro de Investigaciones Medicas Mar Del Plata, Mar del Plata
- Australia (5):
  - Genesiscare North Shore Oncology, St Leonards, New South Wales
  - Blacktown Hospital, Blacktown
  - St Vincent'S Hospital Sydney, Mount Kuring-Gai
  - St John of God Subiaco Hospital, Subiaco
  - Princess Alexandra Hospital, Woolloongabba
- Belgium (5):
  - Cliniques Universitaires Saint-Luc, Brussels
  - Grand Hospital de Charleroi, Charleroi
  - Universitair Ziekenhuis Gent, Ghent
  - Uz Leuven, Leuven
  - Chu de Liă Ge, Liège
- Brazil (5):
  - Hospital de Câncer de Barretos - Fundação Pio XII, Barretos
  - Cepon - Centro de Pesquisas Oncolă"Gicas de Santa Catarina, Florianópolis
  - Centro de Pesquisas Clinicas da Fundação Doutor Amaral Carvalho, Jaú
  - Hospital de Clínicas de Porto Alegre, Porto Alegre
  - Hospital São Lucas Da Pucrs, Porto Alegre
- Chile (5):
  - Biocenter, Concepción
  - Ic La Serena Research, La Serena
  - Centro Del Cancer UC, Santiago
  - Clinica Redsalud Vitacura, Santiago
  - James Lind Centro de Investigacion Del Cancer, Temuco
- France (11):
  - Centre Léon Bérard, Lyon, Rhone
  - Chu Besançon - Hôpital Jean Minjoz, Besançon
  - Hopital Saint Andre, Bordeaux
  - Institut Bergonié, Bordeaux
  - Centre Georges François Leclerc, Dijon
  - Institut Régional Du Cancer de Montpellier, Montpellier
  - Institut Curie - Site de Paris, Paris
  - CRLCC Eugene Marquis, Rennes
  - Ico - Site René Gauducheau, Saint-Herblain
  - Institut Claudius Regaud, Toulouse
  - Institut Gustave Roussy, Villejuif
- Germany (8):
  - Charită - Campus Charită Mitte, Berlin
  - Vivantes Klinikum Neukoelln, Berlin
  - Staedtisches Klinikum Dresden Standort Dresden-Friedrichstadt, Dresden
  - Universitaetsklinikum Heidelberg, Heidelberg
  - Slk-Kliniken Heilbronn Gmbh, Heilbronn
  - Universitäres Krebszentrum Leipzig UCCL, UKL AöR, Leipzig
  - Univ der Johannes GutenbergU, Mainz
  - Universitätsklinikum Münster, Medizinische Klinik A, Münster
- Ireland (5):
  - Cork University Hospital, Cork
  - Mater Misericordiae University Hospital, Dublin
  - Tallaght University Hospital, Dublin
  - St Vincent'S University Hospital, Dublin
  - University Hospital Galway, Galway
- Italy (6):
  - Fondazione Del Piemonte Per L'Oncologia Irccs Candiolo, Candiolo
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - Azienda Socio Sanitaria Territoriale Niguarda (Grande Ospedale Metropolitano Niguarda), Milan
  - Istituto Nazionale Tumori Fondazione G. Pascale, Napoli
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome
  - Istituto Clinico Humanitas, Rozzano
- Japan (8):
  - National Cancer Center Hospital, Chūōku
  - National Cancer Center Hospital East, Kashiwa
  - The Cancer Institute Hospital of Jfcr, Kōtoku
  - National Hospital Organization Shikoku Cancer Center, Matsuyama
  - Shizuoka Cancer Center, Nagaizumi-cho
  - Aichi Cancer Center Hospital, Nagoya
  - Kindai University Hospital, Ōsaka-sayama
  - Saitama Cancer Center, Saitama
- Mexico (3):
  - Medical Care & Research Sa de Cv, Mérida
  - Centro de Atenciă"N E Investigaciă"N Clă Nica En Oncologă A, Mérida
  - Cryptex Investigacion Clinica S.A. de C.V., México
- Netherlands (5):
  - Amsterdam Umc, Locatie Vumc, Amsterdam
  - Universitair Medisch Centrum Groningen, Groningen
  - Radboudumc Nijmegen, Nijmegen
  - Erasmus Medisch Centrum, Rotterdam
  - Umc Utrecht, Utrecht
- Poland (5):
  - SPZOZ Szpital Uniwer w Krakowie, Krakow
  - Instytut MSF Sp. z o.o., Lodz
  - MRUK-MED i Spółka z ograniczoną odpowiedzialnością, Rzeszów
  - Mazowiecki Szpital Wojewodzki W Siedlcach Sp Z O O, Siedlce
  - Aidport Sp Z O.O., Skorzewo
- Portugal (5):
  - Instituto Portuguă S de Oncologia de Lisboa Francisco Gentil, Epe, Lisbon
  - Fundação Champalimaud, Lisbon
  - Centro Hospitalar Universitário de Lisboa Norte, Lisbon
  - Centro Hospitalar Universitario de Santo Antonio, Porto
  - Inst Portude Onco do Porto, Porto
- Spain (8):
  - Hospital Clinic de Barcelona, Barcelona
  - ICO l'Hospitalet - Hospital Duran i Reynals, Barcelona
  - Hospital Universitari Vall D'Hebron, Barcelona
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Virgen Macarena, Seville
- Taiwan (6):
  - China Medical University Hospital, Taichung
  - National Cheng Kung University Hospitalx, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Koo Foundation Sun Yat-Sen cancer center, Taipei
  - Tri-Service General Hospital, Taipei
- Turkey (Türkiye) (6):
  - Gulhane Training and Research Hospital, Ankara
  - Gazi University Medical Faculty, Ankara
  - Ankara University Cebeci Hospital, Ankara
  - Ankara City Hospital, Ankara
  - Medipol Mega University Hospital, Istanbul
  - Izmir Medicalpark Hospital, Izmir

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) on completed studies and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Completed studies that has reached a global end or completion with all data set collected and analyzed, and for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents on completed clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/